CLINICAL TRIAL: NCT03475966
Title: Improving Outcomes in Patients With Hepatobiliary and Pancreatic Cancers With a Nutritional and Physical Conditioning Prehabilitation Program
Brief Title: Improving Outcomes in Cancer Patients With a Nutritional and Physical Conditioning Prehabilitation Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Dr. Franco Carli (Unknown)
Responsible Party: Principal Investigator, Antonio Vigano, Attending Physician, Supportive and Palliative Care Division; Director, Cancer Rehabilitation (CARE) Program; Director, McGill Nutrition and Performance Laboratory, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: prehab_pilot
Record Dates: First submitted 2017-02-28; First posted 2018-03-23 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer; Liver Cancer; Bile Duct Cancer; Hepatobiliary Cancer; Surgery
Keywords: Nutrition; Exercise; Relaxation techniques; Prehabilitation
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Bile Duct Neoplasms; Motor Activity | interventions — Exercise; Nutritional Status; Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Exercise, nutrition and relaxation techniques all beginning four weeks prior to surgery date.
  Interventions: Other: Exercise; Other: Nutrition; Behavioral: Relaxation techniques
- Rehabilitation (Active Comparator): Exercise, nutrition and relaxation techniques all beginning immediately after surgery.
  Interventions: Other: Exercise; Other: Nutrition; Behavioral: Relaxation techniques

INTERVENTIONS:
Other: Exercise — A kinesiologist will provide each patient wih an individualized home-based exercise program including aerobic, resistance and stretching exercises. Patients will also exercise at our clinic once per week under the supervision of the kinesiologist (prehabilitation arm only)
Other: Nutrition — Patients will be asked to fill in a 3-day food diary. A registered dietitian (RD) will review this diary, provide a full nutritional assessment, and ensure patients are following a high-protein diet (1.5 g of protein/kg/day). A whey-protein supplement may be provided to patients, should they require it. The RD will also ensure adequate calorie consumption for weight maintenance and will provided advice to help ease any GI issues the patients may be experiencing.
Behavioral: Relaxation techniques — Patients will see a psychologist who will provide relaxation techniques (eg. imagery, visualization, deep breathing exercises) to help patients manage anxiety prior to surgery.

SUMMARY:
Major surgery is a stressful procedure; good recovery after surgery is important to patients and their doctors. Studies done at the McGill University Health Centre (MUHC) with cancer patients awaiting surgery have shown that exercise combined with simple diet recommendations (which may include a supplement) and relaxation techniques before surgery helped speed up the ability to resume walking after surgery.

These results have made the investigators aware that exercise and good nutrition are as important before surgery as they are after surgery; while it is common practice to start strengthening the body after surgery (rehabilitation), there may be some advantage to begin this process before surgery (prehabilitation).

The purpose of this study is to see if the following program, either before or after surgery, can help patients recover from liver, pancreas or bile duct surgery:

1. Exercise that may help participants move and breath better,
2. Nutrition advice and a supplement to make participants strong,
3. Relaxation and anti-anxiety tips to help cope with the stress of upcoming surgery

The investigators will see if following this program will have an effect on participants' ability to walk before and after surgery.

ELIGIBILITY:
Inclusion criteria:

* A diagnosis or suspicion of either hepatobiliary or pancreatic cancer (primary or metastatic)
* Must be scheduled for surgical resection between 4-6 weeks of recruitment

Exclusion criteria:

* Persons with American Society of Anesthesiologists (ASA) health status class 4-5
* Comorbid medical, physical and mental conditions (eg: dementia, disabling orthopedic and neuromuscular disease, psychosis)
* Cardiac abnormalities
* Severe end-organ disease such as cardiac failure, chronic obstructive pulmonary failure and hepatic failure (alanine aminotransferase and aspartate aminotransferase >50% over the normal range)
* Sepsis
* Morbid obesity (BMI >40)
* Anemia (hematocrit <30 %)
* Other conditions interfering with the ability to perform exercise at home or to complete the testing procedures
* Poor English or French comprehension

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in functional walking capacity as measured by the six-minute walk test (6MWT) | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 meter stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk; encouragement and feedback are given according to published guidelines. They are allowed to rest during the test if needed, but this time is included in the 6 minutes. Reference equations are available for calculating percent of age- and gender-specific norm.

SECONDARY OUTCOMES:
Timed up and go test | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Investigators will measure the time required for a participant to stand up from being seated, walk a distance of 3 metres, turn around and walk back to the chair, and sit down. This measure will be administered based on Canadian Society for Exercise Physiology standards.
30-second sit to stand test | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Investigators will measure the number of times participants can stand from a seated position in 30-seconds. This measure will be administered based on Canadian Society for Exercise Physiology standards.
30-second arm curl test | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Investigators will measure the number of times participants can perform a full arm curl in 30-seconds. Both arms will be assessed, one at a time. This measure will be administered based on Canadian Society for Exercise Physiology standards.
Change in handgrip strength | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  To be measured using the Jamar hydraulic hand dynamometer. Two measures from each hand will be taken, with patient seated and arm bent at a 90-degree angle. The average of the two measures for each hand will be recorded and compared to normative data.
Change in body composition | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Body composition will be measured via dual-energy X-ray absorptiometry (DXA; Lunar Prodigy Advance, General Electric Healthcare, Madison, WI). Studies from the McGill Nutrition and Performance Laboratory group have validated the use of DXA in advanced cancer patients.
Assessment of food intake and change over study period | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Participants will be asked to bring a 3-day food diary to their baseline visit to obtain detailed information about the quantity and type of food and beverages consumed during a non-consecutive 3-day period. Overall energy intake, as well as macronutrient distribution (e.g., amount of carbohydrates, fats, proteins, and fibre at each meal) will be calculated using the Food Processor SQL Nutrition Analysis software.
Perioperative data | 7 days post-operatively
  This data will include operative characteristics, transfusion rates, length of surgery, intraoperative complications and length of stay.
Postoperative complications | 4 weeks post-operatively
  Including surgical site infection, other infectious complications (such as pneumonia, urinary tract infection, line sepsis), bile leak, hemorrhage, deep vein thrombosis, etc., will be recorded and scored using the Clavien Classification.
Health-related quality of life (HRQL) - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  As measured by the acute (1 week recall period) Functional Assessment of Cancer Therapy (FACT) survey. This questionnaire also has versions that identify symptoms more specific to hepatobiliary and colorectal cancer patients; this is of relevance to this study given liver metastasis occurs in these patients. The questionnaire is separated into five subscales: 1) physical well-being, 2) social/family well-being, 3) emotional well-being, 4) functional well-being, 5) additional concerns (specific to cancer type). Each question is scored 0-4 on a likert scale, with 0 indicating, "not at all," and 4 indicating, "very much." These scores are then reversed where applicable and added. A higher score indicates better QoL.
The Edmonton Symptom Assessment System (ESAS) - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Currently used at the MUHC Cedars Cancer Centre to assist in the assessment of pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath. Each symptom is rated from 0 to 10 on a numerical scale based on severity, with 0 indicating that the symptom is absent and 10 that it is the worst possible severity.
Physical activity level - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire. The CHAMPS is a self-reported measure of physical activity, comprising 41 activities evaluated according to the total number of hours done during an average week. Each physical activity is assigned a metabolic equivalent (MET) value yielding average weekly caloric expenditure for the listed physical activities. There is evidence for the validity of CHAMPS as a measure of postoperative recovery. Data will be categorized as either mild, moderate or intense activity and changes in the number of hours spent performing activities within each category will be assessed.
Nutritional status - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  To be assessed using the Abridged Patient-Generated Subjective Global Assessment (aPG-SGA); a validated questionnaire used to assess the nutritional and functional status of cancer patients. The scoring system allows patients at risk for malnutrition to be identified and triaged for nutritional intervention. The aPG-SGA may also be useful in monitoring short-term changes in nutritional status. A score ≥9 indicates a critical need for nutritional intervention.
Fatigue - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  To be assessed using a visual analog scale (1-10) and the Brief Fatigue Inventory (BFI). The BFI assesses the level of fatigue and its impact on activities of daily living. The test has 9 questions: three questions are designed to assess the patient's fatigue during the immediate waking hours and 6 questions address how fatigue has interfered in the patient's life over the previous 24 hours. Each question uses a scale rating from "0" (no fatigue) to "10" (unimaginable fatigue) for a total of 90 points.
Weight - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Body weight will be measured (Kg)
Height | Baseline
  Height will be measured with a stadiometer (m)
Body mass index - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Calculated wt (kg)/ht^2 (m)
Blood pressure - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Systolic and diastolic at rest (mmHg)
Heart rate - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Beats per minute measured using a pulse oximeter

OTHER OUTCOMES:
Lower extremity strength - assessment of change over time | Baseline, pre-operative assessment, 4 weeks post-operative, 8 weeks post-operative
  Optional measure: assessed using the Biodex System 3 (Biodex Medical Systems, Shirley, NY).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Vigano, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No